CLINICAL TRIAL: NCT03527823
Title: The Comparison of Granulosa Cell Apoptosis Rates on Microdose Flare up GnRH Analog Protocol Versus Luteinizing Hormone Administrated Microdose Flare up GnRH Analog Protocol in Poor Ovarian Responders Undergoing in Vitro Fertilization.
Brief Title: The Comparison of Granulosa Cell Apoptosis Rates With or Without Luteinizing Hormone Administration in Poor Responders.
Status: Completed | Type: Observational
Sponsor: Sebnem Alanya Tosun (Other)
Collaborators: Giresun University Funding for Scientific Research Project (Unknown)
Responsible Party: Sponsor-Investigator, Sebnem Alanya Tosun, Assistant Professor- Obstetrics and Gynaecology, Giresun University
Organization: Giresun University (Other)
Other Study IDs: GranulosaApoptosis; 123 (Other: Giresun University Scientific Research Project)
Record Dates: First submitted 2018-04-25; First posted 2018-05-17 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Fertilization in Vitro
Keywords: Fertilization in Vitro; Granulosa Cells; Apoptosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — folicular aspiration fluid sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LH supplementation: luteinizing hormone administrated microdose flare up GnRH analog protocol in poor ovarian responders undergoing in vitro fertilization.
- without LH supplementation: microdose flare up GnRH analog protocol in poor ovarian responders

SUMMARY:
In Zeynep Kamil Women and Children's Education and Research Hospital which is a tertiary referral hospital, the investigators perform microdose flare-up gonadotropin-releasing hormone (GNRH) analogue or GNRH antagonist protocol to the poor responders. The investigators may or may not supplement luteinizing hormone (LH). Human chorionic gonadotropin (hCG) triggering is performed when at least 2 follicles diameter are above 17 mm and the serum estradiol level is above 500 pg / ml. 36 hours after hCG, ovarian aspiration is performed by the guidance of transvaginal ultrasound. Normally after oocyte separation process, the remaining follicle aspiration fluid is destroyed.

n the present study, the follicle aspiration fluid is planned to be used with the patient's permission. The investigators are going to examine the granulosa cell apoptosis rate by using annexin-5 antibody in both groups 1 (LH added) and 2 (without LH).

For this purpose, a total of 40 volunteer patients are planned to involve, the groups are designed as 20 LH added and 20 LH added women.

In the present study, the investigators hypothesis that the rates of granulosa cell apoptosis in poor responders may be different between the group 1 (with LH) and group 2 (without LH), this will lead to IVF therapy in the near future.

DETAILED DESCRIPTION:
The supplementation of human menopausal gonadotropin (HMG) in terms of luteinizing hormone (LH) support in controlled ovarian stimulation (COS) is a controversial issue. Follicle stimulating hormone (FSH) and LH are required for ovarian steroidogenesis in anovulatory women with gonadotropin deficiency according to the two cell-two gonadotropin hypothesis. LH supplementation is needed to ensure adequate follicular estradiol (E2) production during the follicular phase, completion of oocyte maturation and development in the endometrium. Despite, the need for LH for ovarian stimulation in normogonadotropic women is controversial. Additional LH supplementation during stimulation with FSH may provide an advantage in increasing follicle development and thus may be shortening the duration of treatment. It has been suggested that the change of gonadotropins from FSH to LH in the presence of ovarian stimulation is beneficial in the development of a more homogeneous follicular cohort [1] [2]. However, contrary opinions have reported that LH supplementation does not bring any additional benefit [3].

In recent years, studies have been done to investigate the utility of the addition of LH as well as FSH to the cycle outcome. In a Cochrane review, the combination of recombinant follicle stimulating hormone (r-FSH) and recombinant luteinizing hormone (r-LH) administration in in vitro fertilization/intracytoplasmic sperm injection (IVF / ICSI) cycles compared to only r-FSH cycles in 14 randomized controlled trials [4]. When r-LH was added, there was no statistical difference in terms of pregnancy outcomes. However, due to the small size of the work, the net result was not achieved. The other study supported the treatment of rFSH alone, while the addition of r-LH was found to be beneficial only in one of the studies [5, 6] . As a result, there is no significant difference in live birth rates.

However, the studies in only poor responders showed a significant increase in pregnancy rates with the addition of r-LH [5, 7]. In contrast, recently Bosch et al. reported that the addition of r-LH in the 36-39 age group of patients with GnRH antagonist protocol benefit from LH support, while patients under the age of 36 do not [8]. In conclusion, there is no consensus to administrate r-LH to the protocols of poor responders. Our hypothesis is LH administration may decrease granulosa apoptosis rate in follicular fluids and may be beneficial to poor responders and over age of 35.

In Zeynep Kamil Women and Children's Education and Research Hospital where the data of study patients is going to be collected, the investigators are applying microdose flare-up GNRH analogue or GNRH antagonist protocol to the poor responders. The investigators may or may not supplement LH. hCG is performed when at least 2 follicles are 17 mm and the serum estradiol level is above 500 pg / ml. 36 hours after hCG, ovarian aspiration is performed by the guidance of transvaginal ultrasound. Normally after oocyte separation process, the remaining follicle aspiration fluid is destroyed.

The follicle aspiration fluid is planned to be used within the permission of the patient in the present study. The investigators are going to examine the granulosa cell apoptosis rate with using annexin-5 antibody in group 1 (LH added) and group 2 (without LH).

For this purpose, a total of 40 volunteer patients are planned to have 20 LH added and 20 LH added patient groups.

Statistical analysis is going to be performed using SPSS 11 program. p <0.05 will be considered significant.

In the present study, the investigators hypothesis that comparing the rates of granulosa cell apoptosis in poor responders as two different groups (with and without addition of LH) will lead to IVF therapy in the near future.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 aged female
* poor ovarian responders
* undergoing treatment for primary/secondary infertility

Exclusion Criteria:

* endocrinologic or metabolic disorders

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female population in reproductive age undergoing infertility treatment
Study Population: 18-49 aged females who undergoes IVF treatment and who are defined as poor responders
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
the comparison of granulosa cell apoptosis rate with or without LH supplementation in poor responders | June 2018-August 2018
  the investigators hypothesized that granulosa cell apoptosis rate on luteinizing hormone supplemented microdose flare up GnRH analog protocol in poor ovarian responders undergoing in vitro fertilization would be lower than not administered protocol

CONTACTS AND LOCATIONS:
Overall Officials: enis ozkaya, Study Director — zeynep kamil education and research hospital
Locations (1):
- Sebnem Alanya Tosun, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bosch E, Labarta E, Crespo J, Simon C, Remohi J, Pellicer A. Impact of luteinizing hormone administration on gonadotropin-releasing hormone antagonist cycles: an age-adjusted analysis. Fertil Steril. 2011 Mar 1;95(3):1031-6. doi: 10.1016/j.fertnstert.2010.10.021. Epub 2010 Nov 10. PMID 21067717
- [Background] Ferraretti AP, Gianaroli L, Magli MC, D'angelo A, Farfalli V, Montanaro N. Exogenous luteinizing hormone in controlled ovarian hyperstimulation for assisted reproduction techniques. Fertil Steril. 2004 Dec;82(6):1521-6. doi: 10.1016/j.fertnstert.2004.06.041. PMID 15589853
- [Background] Kaleli S, Yanikkaya-Demirel G, Erel CT, Senturk LM, Topcuoglu A, Irez T. High rate of aneuploidy in luteinized granulosa cells obtained from follicular fluid in women who underwent controlled ovarian hyperstimulation. Fertil Steril. 2005 Sep;84(3):802-4. doi: 10.1016/j.fertnstert.2005.02.040. PMID 16169431
- [Background] Sullivan MW, Stewart-Akers A, Krasnow JS, Berga SL, Zeleznik AJ. Ovarian responses in women to recombinant follicle-stimulating hormone and luteinizing hormone (LH): a role for LH in the final stages of follicular maturation. J Clin Endocrinol Metab. 1999 Jan;84(1):228-32. doi: 10.1210/jcem.84.1.5389. PMID 9920089
- [Background] Filicori M, Cognigni GE, Samara A, Melappioni S, Perri T, Cantelli B, Parmegiani L, Pelusi G, DeAloysio D. The use of LH activity to drive folliculogenesis: exploring uncharted territories in ovulation induction. Hum Reprod Update. 2002 Nov-Dec;8(6):543-57. doi: 10.1093/humupd/8.6.543. PMID 12498424
- [Background] Balasch J, Vidal E, Penarrubia J, Casamitjana R, Carmona F, Creus M, Fabregues F, Vanrell JA. Suppression of LH during ovarian stimulation: analysing threshold values and effects on ovarian response and the outcome of assisted reproduction in down-regulated women stimulated with recombinant FSH. Hum Reprod. 2001 Aug;16(8):1636-43. doi: 10.1093/humrep/16.8.1636. PMID 11473955
- [Background] Mochtar MH, Van der Veen, Ziech M, van Wely M. Recombinant Luteinizing Hormone (rLH) for controlled ovarian hyperstimulation in assisted reproductive cycles. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD005070. doi: 10.1002/14651858.CD005070.pub2. PMID 17443569
- [Background] Tarlatzis B, Tavmergen E, Szamatowicz M, Barash A, Amit A, Levitas E, Shoham Z. The use of recombinant human LH (lutropin alfa) in the late stimulation phase of assisted reproduction cycles: a double-blind, randomized, prospective study. Hum Reprod. 2006 Jan;21(1):90-4. doi: 10.1093/humrep/dei293. Epub 2005 Sep 19. PMID 16172149
- [Background] De Placido G, Alviggi C, Perino A, Strina I, Lisi F, Fasolino A, De Palo R, Ranieri A, Colacurci N, Mollo A; Italian Collaborative Group on Recombinant Human Luteinizing Hormone. Recombinant human LH supplementation versus recombinant human FSH (rFSH) step-up protocol during controlled ovarian stimulation in normogonadotrophic women with initial inadequate ovarian response to rFSH. A multicentre, prospective, randomized controlled trial. Hum Reprod. 2005 Feb;20(2):390-6. doi: 10.1093/humrep/deh625. Epub 2004 Dec 2. PMID 15576390